CLINICAL TRIAL: NCT02714816
Title: Natural History Study of Patients With Leber Congenital Amaurosis Associated With Mutations in RPE65
Status: Completed | Type: Observational
Sponsor: MeiraGTx UK II Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: MGT005
Record Dates: First submitted 2016-03-08; First posted 2016-03-22 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Leber Congenital Amaurosis
MeSH Terms: conditions — Leber Congenital Amaurosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
MGT005 is a natural history study to collect longitudinal prospective data from patients with Leber Congenital Amaurosis associated with defects in RPE65.

DETAILED DESCRIPTION:
Leber Congenital Amaurosis (LCA) is a diagnosis for a group of severe, autosomal recessively inherited rod - cone dystrophies that typically result in complete visual loss in the third or fourth decade of life. One form, LCA2, is caused by a mutation in the gene encoding RPE56, an RPE-specific 65-kDa isomerase. Non-functional RPE65 results in photoreceptor cells that are unable to respond to light resulting in these patients being visually impaired.

In preparation for human clinical trials, a detailed prospective phenotypic study will be undertaken to investigate the natural history of RPE65-LCA. Such a study will help identify suitable patients for therapeutic intervention. Furthermore through greater phenotyping an optimal window for intervention and specific parameters to help quantify effect and identify clinical end points may have been ascertained .

ELIGIBILITY:
Inclusion Criteria:

* Patients with RPE65 associated retinal dystrophy
* Minimum subject age of 3 years
* Able to give consent/parent or guardian able to give consent

Exclusion Criteria:

* Patients unable or unwilling to undertake consent or clinical testing
* Have received a gene therapy treatment in both eyes

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with RPE65-LCA condition
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2016-04; Primary Completion 2023-07-22 (Actual); Study Completion 2023-07-22 (Actual)

PRIMARY OUTCOMES:
Analysis of retinal structure and function | 6 years
  Retinal structure will be analysed using Adaptive optics and SD-OCT and Fundal autofluorescence. This will be correlated with assessment of visual acuity, psychophysical visual assessment, visual mobility, retinal sensitivity and visual fields

SECONDARY OUTCOMES:
Quality of Life Questionnaires | 6 years
  Assessment of Visual impairment using appropriate, validated questionnaires
Retinal Sensitivity | 6 years
  To be assessed in Microperimetry
Retinal Structural analysis | 6 years
  Retinal Structure analysis with Adaptive Optics
Fundal Autofluorescence | 6 years
  Presence or Absence
Assessment of Visual Fields | 6 years
  Assessment of Visual Fields with analysis of hill of vision

CONTACTS AND LOCATIONS:
Overall Officials: Michel Michealides, Prof, Principal Investigator — UCL/Moorfileds
Locations (2):
- Kellogg Eye Center, Ann Arbor, Michigan, United States
- Moorfields Eye Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kumaran N, Georgiou M, Bainbridge JWB, Bertelsen M, Larsen M, Blanco-Kelly F, Ayuso C, Tran HV, Munier FL, Kalitzeos A, Michaelides M. Retinal Structure in RPE65-Associated Retinal Dystrophy. Invest Ophthalmol Vis Sci. 2020 Apr 9;61(4):47. doi: 10.1167/iovs.61.4.47. PMID 32347917
- [Derived] Kumaran N, Rubin GS, Kalitzeos A, Fujinami K, Bainbridge JWB, Weleber RG, Michaelides M. A Cross-Sectional and Longitudinal Study of Retinal Sensitivity in RPE65-Associated Leber Congenital Amaurosis. Invest Ophthalmol Vis Sci. 2018 Jul 2;59(8):3330-3339. doi: 10.1167/iovs.18-23873. PMID 30025081